CLINICAL TRIAL: NCT07199335
Title: A Multi-Center Assessment of an Intervention to Provide Long-Acting Cabotegravir Injectable Pre-Exposure Prophylaxis to People Who Inject Drugs
Brief Title: Long-acting Cabotegravir Injectable Pre-exposure Prophylaxis for People Who Inject Drugs
Acronym: ASCEND
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ViiV Healthcare (Industry); Fenway Community Health (Other)
Responsible Party: Principal Investigator, Suzanne McCluskey, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025P002398
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: HIV; Substance Use Disorder (SUD); Injection Drug Use
Keywords: HIV; Substance use; pre-exposure prophylaxis; cabotegravir; long-acting cabotegravir; PrEP; implementation science; PrEP navigator
MeSH Terms: conditions — Substance-Related Disorders | interventions — cabotegravir

STUDY DESIGN:
Intervention Model Description: This is an implementation study, using long-acting injectable cabotegravir for its approved indication as HIV pre-exposure prophylaxis for people with sexual risk factors for HIV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All participants (Experimental): All participants will receive long-acting injectable cabotegravir and a suite of support services, including PrEP navigation, transportation assistance, and financial incentives.
  Interventions: Drug: APRETUDE (cabotegravir)

INTERVENTIONS:
Drug: APRETUDE (cabotegravir) — All participants will be prescribed APRETUDE based on APRETUDE's FDA approved indication, which is sexual risk of HIV transmission.

SUMMARY:
The goal of this study is to determine the feasibility and impact of delivering long-acting injectable cabotegravir HIV pre-exposure prophylaxis and suite of support services to adults who inject non-prescription drugs who are risk for HIV through known sexual risk.

DETAILED DESCRIPTION:
This is a Phase IV open-label single arm implementation study of the on-label use of an FDA approved drug, cabotegravir, as long-acting, injectable HIV pre-exposure prophylaxis (CAB-LA) among people who inject drugs. All enrollees will be prescribed CAB-LA based on CAB-LA's FDA approved indication, which is sexual risk of HIV transmission. Investigators will recruit participants from two sites in Boston, Massachusetts. The target study sample size is 100 participants.

Recruitment will be primarily by clinician referrals and medical records review at each site.

The study team will screen potential participants at both sites and assess their initial eligibility. Participants will be eligible to participate if they meet the inclusion and exclusion criteria. If an individual consents to participation, a 4th generation antibody/antigen (Ab/Ag) screening test (rapid or lab-based) and a confirmatory HIV-1 RNA test will be sent. If the HIV Ab/Ag screening test is negative, individuals will be enrolled.

Once a participant is enrolled, the participant will return 0-7 days later to complete a medical evaluation by a medical provider who will prescribe CAB-LA, and the participant will complete an enrollment survey. After the enrollment survey, participants will receive the first CAB-LA injection according to label instructions. The second injection visit will occur 1 month after the first injection. Thereafter, CAB-LA will be administered every 2 months for three additional doses. Thus, participants will remain in the study for seven months. CAB-LA for the study is supplied by ViiV Healthcare Ltd.

At each CAB-LA injection visit after the first one, participants will be asked to complete a short survey. A longer survey will be administered at the final study visit for each participant regarding acceptability of the intervention.

At each follow-up study visit prior to CAB-LA injection, HIV testing will be performed using both a screening Ag/Ab test and a confirmatory HIV-1 RNA test (if a blood sample for RNA testing can be obtained). If the screening HIV Ag/Ab test is positive, the CAB-LA injection will not be administered, and the participant will be withdrawn from the study and referred for HIV treatment. If the confirmatory HIV-1 RNA test returns positive from any study visit, including from the pre-enrollment sample, the participant will be withdrawn from the study and referred for HIV treatment. For any participant who is diagnosed with HIV during the study period, additional testing for antiretroviral drug resistance, including integrase strand transfer inhibitor resistance, will be collected, and the patient will be referred to HIV care.

Participants will also be screened for STIs (gonorrhea, chlamydia, and syphilis), HBV, and HCV at enrollment and at the time of the 3rd and 5th injections.

In addition to receiving CAB-LA, each participant will also receive support services while participating in the study. Specifically, participants will be connected with a PrEP Navigator who will work with participants between visits to provide support, education, and coordinate visits. The PrEP navigator will be a trained non-provider who can provide counseling about the risks and benefits of PrEP, discuss participant concerns, assist in coordinating clinic visits, and facilitate connections to medical care if needed. In addition, incentives for phlebotomy ($20) and appointment attendance ($20) will be provided to all participants. Transportation assistance for study appointments will also be provided.

After the study, participants will transition from study-supplied CAB-LA to commercially-available CAB-LA.

ELIGIBILITY:
Inclusion Criteria:

* HIV Ab/Ag test (lab-based or rapid) negative at time of enrollment
* ≥18 years old
* Able to provide informed consent
* Have injected non-prescribed drugs within the past 6 months
* No prior history of receiving cabotegravir (Note: prior or active use of non-CAB PrEP ([FTC/TDF or FTC/TAF]) at screening is allowed, but participant will need to indicate that they prefer to switch to injectable PrEP).
* PrEP provider deems cabotegravir use to be appropriate per the applicable prescribing information prior to enrollment in the study.

Exclusion Criteria:

* Pregnant or breastfeeding people. Should a participant become pregnant, the treating physician will discuss with the participant whether to continue study medication, taking into consideration the risks and benefits of continuing cabotegravir compared with the risk of switching to an alternative recommended PrEP regimen.
* Has not had vaginal or anal sex in the past 6 months
* HIV indeterminate or positive test result during screening and prior to initiation of CAB PrEP
* Already diagnosed with HIV
* Taking any of the following medications: Carbamazepine, Rifampin, Oxcarbazepine, Rifapentine, Phenobarbital, Phenytoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Persistence on CAB-LA | 7 months
  For the primary analysis, investigators will calculate the proportion of study participants who achieve PrEP persistence at 7 months post-initiation. Investigators will then calculate 95% confidence intervals around the proportion.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fenway Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
IPD will not be shared publicly. IPD can be made available upon request to the principal investigator with proof of IRB approval and a fully executed data use agreement.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data can be made available upon request following completion of study.
Access Criteria: IPD can be made available upon request to the principal investigator with proof of IRB approval and a fully executed data use agreement.